CLINICAL TRIAL: NCT00003345
Title: Phase II Trial of Cisplatin and Irinotecan in Patients With Suboptimally Debulked, Incompletely Responding Ovarian Cancer
Brief Title: Cisplatin Plus Irinotecan in Treating Patients With Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-121; CDR0000066322 (Registry Identifier: PDQ (Physician Data Query)); NCI-H98-0013
Record Dates: First submitted 1999-11-01; First posted 2004-03-30 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; Irinotecan

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining cisplatin and irinotecan in treating patients who have ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antitumor effect of weekly cisplatin and irinotecan in patients with suboptimally debulked ovarian, fallopian tube, or peritoneal cancer and persistently elevated serum values of CA125 after 3 courses of standard therapy with paclitaxel and either carboplatin or cisplatin. II. Evaluate the toxicity, both qualitative and quantitative, of this regimen in this patient population. III. Evaluate the quality of life of these patients.

OUTLINE: Patients receive cisplatin IV over 30 minutes followed by irinotecan IV over 90 minutes. Treatment is administered weekly for 4 weeks (days 1, 8, 15, and 22) followed by 2 weeks of rest. Patients receive at least 3 courses (18 weeks) of therapy in the absence of disease progression or unacceptable toxicity. If patients demonstrate complete response to treatment, they are encouraged to undergo second-look laparoscopy or laparotomy. Quality of life is assessed before treatment, after the first course, and then after every 2 courses of therapy. Patients are followed 30 days after the last treatment and then for survival.

PROJECTED ACCRUAL: There will be 12-35 patients accrued into this study over 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed epithelial carcinoma of the ovary, fallopian tube, or peritoneum At least 3 prior courses of standard platinum-paclitaxel regimen Patients with taxane allergy may enter this study after 3 courses of platinum based treatment CA125 at least 35 measured within 30 days of commencement of treatment Measurable disease not required No CNS metastases, carcinomatous meningitis or interstitial pulmonary fibrosis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Calcium less than 12.0 mg/dL Cardiovascular: No unstable angina No New York Heart Association grade III or IV cardiac disease Pulmonary: See Disease Characteristics Other: No active or uncontrolled infection No history of seizures No known Gilbert's Disease No medical or psychiatric conditions that makes patient a poor risk for participation in this study Not pregnant or lactating Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior irinotecan or topotecan Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the pelvis Surgery: At least 4 weeks since prior surgery and recovered Other: No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1997-10; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States